CLINICAL TRIAL: NCT06930742
Title: Mindfulness-Enhanced Cognitive-Motor Dual-Task Training Using Balance and Isokinetic Systems for Parkinson's Disease With Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: Mindfulness-Enhanced Dual-Task Training in PD-MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Mingzhou Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jingzhi Zhang, technician in charge, Nanjing Mingzhou Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NJKF202503001
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment (MCI); Parkinson's Disease (PD)
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MDT group (Experimental): Mindfulness-enhanced Dual-task Training
  Interventions: Device: Cognitive-Motor Dual-Task Training; Other: Mindfulness Training
- DT group (Active Comparator): Dual-task Training
  Interventions: Device: Cognitive-Motor Dual-Task Training; Other: Quiet Rest
- ST group (Active Comparator): Single-task Training
  Interventions: Device: Single-task Training; Other: Quiet Rest

INTERVENTIONS:
Device: Cognitive-Motor Dual-Task Training — Participants perform physical exercises using the balance training system and isokinetic muscle strength training system while simultaneously completing cognitive tasks to improve motor-cognitive coordination. The training follows a task-segmentation approach:
  Balance Task Module: Participants perform dynamic balance training on the balance training system while engaging in cognitive tasks (e.g., digit span, arithmetic, or word fluency tasks).
  Strength Task Module: Participants conduct isokinetic strength training while performing corresponding cognitive tasks.
  Task difficulty is progressively adjusted based on participant performance.
  Arms: DT group; MDT group
Other: Mindfulness Training — Guided by a professional mindfulness instructor, participants engage in mindfulness meditation to enhance attention, emotional regulation, and cognitive readiness. The training includes breath awareness, body scan, and present-moment awareness, delivered through guided meditation.
  Arms: MDT group
Device: Single-task Training — Participants perform physical exercises using the balance training system and isokinetic muscle strength training system without any concurrent cognitive tasks. The training follows a task-segmentation approach, including dynamic balance training and isokinetic strength training to enhance motor function.
  Arms: ST group
Other: Quiet Rest — Participants remain seated in a quiet environment without engaging in mindfulness training or cognitive tasks.
  Arms: DT group; ST group

SUMMARY:
The goal of this clinical trial is to learn if Mindfulness-Enhanced Dual-Task Training work to treat PD-MCI in adults. The main questions it aims to answer are:

Does Mindfulness-Enhanced Dual-Task Training improve the cognitive or motor function of participants? Can the combination of Dual-Task Training and Mindfulness achieve better effects?

Researchers will compare 3 groups (Dual-Task Training + Mindfulness, Dual-Task Training, and conventional motor task training) to see if Dual-Task Training and Mindfulness works to treat PD-MCI.

Participants will:

Receive treatment for 4 weeks Receive scale and instrument testing before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 55 and 75 years.
* Disease Diagnosis: Clinically diagnosed with Idiopathic Parkinson's Disease (PD) according to the UK Parkinson's Disease Society Brain Bank Criteria.
* Disease Stage: Hoehn & Yahr (H&Y) stages 1 to 2.5.
* Cognitive Function: Montreal Cognitive Assessment (MoCA) score between 23 and 26, indicating mild cognitive impairment (MCI).
* Medication Stability: Stable doses of antiparkinsonian medications for at least 4 weeks prior to screening.
* Subjective Cognitive Complaints: Self-reported or informant-reported cognitive decline persisting for at least 6 months.
* Ambulatory Ability: Able to walk independently, with or without assistive devices.
* Sensory Abilities: Adequate vision and hearing to comply with study procedures.
* Informed Consent: Willingness to provide written informed consent and comply with study requirements.

Exclusion Criteria:

* Other Neurological Disorders: Presence of other neurological conditions that could affect cognitive function, such as Alzheimer's disease, stroke, or brain tumors.
* Psychiatric Conditions: Severe psychiatric disorders, including major depressive disorder or schizophrenia.
* Substance Abuse: Recent history of drug or alcohol abuse.
* Serious Medical Conditions: Uncontrolled hypertension, diabetes, heart disease, or other conditions that could interfere with study participation or outcomes.
* Severe Cognitive Impairment: Diagnosis of Parkinson's Disease Dementia (PDD).
* Other Factors Affecting Cognition: Recent head trauma, uncontrolled thyroid dysfunction, vitamin B12 deficiency, or other conditions known to affect cognitive function.
* Deep Brain Stimulation (DBS): History of DBS treatment. Participation in Other Clinical Trials: Participation in another clinical trial that could interfere with this study within the last 3 months.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | From enrollment to the end of treatment at 4 weeks
  The Montreal Cognitive Assessment (MoCA) is a widely used neuropsychological tool for detecting mild cognitive impairment (MCI). It assesses multiple cognitive domains, including attention, executive function, memory, language, visuospatial ability, abstraction, calculation, and orientation. The total score is 30 points, with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Mingzhou Rehabilitation Hospital, Nanjing, Jiangsu, China